CLINICAL TRIAL: NCT03011294
Title: Cardiovascular Impact, Quality e Quantity of Sleep in Bed Partners of Patients With Obstructive Sleep Apnea: a Randomized Study
Brief Title: Cardiovascular Impact, Quality e Quantity of Sleep in Bed Partners of Patients With Obstructive Sleep Apnea
Acronym: SLEEP-PARTNERS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Luciano F Drager, MD, PhD, Associate Professor of Medicine, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SDC 4165.14.145
Record Dates: First submitted 2016-12-27; First posted 2017-01-05 (Estimated); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Sleep Apnea Syndromes
MeSH Terms: conditions — Sleep Apnea Syndromes | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CPAP (in the partner) (Active Comparator): Positive airway pressure for treating OSA in the bed partner.
  Interventions: Device: Continuous positive airway pressure (CPAP)
- Nasal strips (in the partner) (Placebo Comparator): Nasal dilator as a placebo for treating OSA in the bed partner.
  Interventions: Device: Nasal strip

INTERVENTIONS:
Device: Continuous positive airway pressure (CPAP) — Standard treatment for sleep apnea
  Arms: CPAP (in the partner)
Device: Nasal strip — Placebo
  Arms: Nasal strips (in the partner)

SUMMARY:
Obstructive sleep apnea (OSA) is a common clinical condition associate with a negative impact not limited to the patients but also to the partner that sleep in the same bed. Is it reasonable to speculate that the partner suffer sleep deprivation, increased level of irritability, insomnia, fatigue, among others due to the loud snoring caused by the OSA patient. Although previous data reported impaired sleep quality in partners of patients with OSA, it is not clear in literature whether OSA promotes cardiovascular impact and if the treatment of OSA promotes some cardiovascular benefits in (the) partner beyond the improvements in the subjective and objective sleep. Thus, the main objectives of this randomized controlled study are: to evaluate the impact of three months of randomization (treatment with nasal CPAP or nasal strips) on the endothelial function, blood pressure (ambulatory blood pressure monitoring), sleep duration (wrist actigraphy for 1 week) and sleep quality (Pittsburgh Questionnaire) and the frequency of OSA in the bed partners of patients with moderate to severe OSA.

ELIGIBILITY:
Inclusion Criteria:

* Bed partners of patients with moderate to severe OSA

Exclusion Criteria:

* Bed partners with OSA using specific treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Endothelial function (forearm dilation, FMD - %) | 3 months

SECONDARY OUTCOMES:
Sleep quantity (measured by actigraphy - hours/night) | 3 months
  1 week of wrist actigraphy
Sleep quality (Pittsburgh Questionnaire) | 3 months
Ambulatory blood pressure monitoring (ABPM) | 3 months
Frequency of OSA | Baseline only

CONTACTS AND LOCATIONS:
Locations (1):
- Luciano Drager, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No